CLINICAL TRIAL: NCT01019174
Title: An Open, Randomized Clinical Phase I/II Trial to Investigate Maximum Tolerated Dose, Efficacy, and Safety of Lenalidomide/Low-dose Dexamethasone in Combination With Continuous Oral Cyclophosphamide Compared to Lenalidomide/Low-dose Dexamethasone Combined With Single Cyclophosphamide Doses IV in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Lenalidomide/Low-dose Dexamethasone in Combination With Continuous Oral Cyclophosphamide Compared to Lenalidomide/Low-dose Dexamethasone Combined With Single Cyclophosphamide Doses IV in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: MM_LEN_DEX_CY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-DSMM-0279; GMIHO-005/2008 (Other: GMIHO)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2014-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral application (Active Comparator): oral application Cyclophosphamide
  Interventions: Drug: Cyclophosphamide
- intravenous application (Active Comparator): intravenous application Cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — comparison of lenalidomide/low-dose dexamethasone in combination with continuous oral cyclophosphamide to lenalidomide/low-dose dexamethasone combined with single cyclophosphamide doses intravenous
  Other Names: Revlimid; Endoxan
  Arms: oral application
Drug: Cyclophosphamide — comparison of lenalidomide/low-dose dexamethasone in combination with continuous oral cyclophosphamide to lenalidomide/low-dose dexamethasone combined with single cyclophosphamide doses intravenous
  Other Names: Revlimid; Endoxan
  Arms: intravenous application

SUMMARY:
The purpose of this study is to investigate the efficacy and tolerability of LEN/low-dose DEX and continuous low-dose CY administered orally compared to LEN in combination with low-dose DEX and single CY doses IV in patients with relapsed MM.

DETAILED DESCRIPTION:
This is an open, randomized, multicenter, phase I/II study with a parallel group design investigating an intravenous and an oral CY dosing schedule in combination with LEN and low-dose DEX in patients with refractory or relapsed MM. In phase I MTD of CY will be determined using a common dose escalation scheme with 3 to 6 patients per dose level. In phase II, efficacy and safety of the treatment regimens at the MTD will be investigated in 20 patients.

ELIGIBILITY:
INCLUSION CRITERIA

1. Understand and voluntarily sign an informed consent form.
2. Age at least 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Previously diagnosed with multiple myeloma based on standard criteria and requires therapy for primary refractory disease or 1st - 3rd relapse because of progressive disease (PD), defined as a 25% increase in M-protein, development of new or worsening of existing lytic bone lesions or soft tissue plasmacytoma, or hypercalcemia (serum calcium > 11.3 mg/dL), or clinical relapse from CR.
5. At least one measurable disease manifestation defined as follows:

   * For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value (generally, but not exclusively, > 1g/dL IgG M-protein or > 0.5 g/dL IgA) and, where applicable, urine light-chain excretion of ≥ 200 mg/24 h.
   * For oligo- or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or a quantifiable plasma cell infiltration of the bone marrow as determined by bone marrow biopsy.
6. ECOG performance status equal to or less than 2 at time of randomization/registration (see Appendix I).
7. Laboratory test results within these ranges within 1 week prior to randomization/registration:

   * Absolute neutrophil count ≥ 1.5 x 109/L without the use of colony stimulating factors within 14 days before the laboratory test.
   * Platelet count ≥ 75 x 109/L without transfusion support within 14 days before the laboratory test.
   * Hemoglobin ≥ 7.5 g/dL (regardless of transfusion support or prior medication with erythropoietin).
   * Calculated creatinine clearance ≥ 50 mL/minute.
   * Total bilirubin equal to or less than 1.5 mg/dL.
   * AST (SGOT) and ALT (SGPT) equal to or less than 2,5 x ULN.
   * Corrected serum calcium < 14 mg/dL (< 3.5 mmol/L).
8. Female subjects of childbearing potential must:

   * Understand that the study medication could have a potential teratogenic risk
   * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception:

     * Implant
     * Levonorgestrel-releasing intrauterine system (IUS)
     * Medroxyprogesterone acetate depot
     * Tubal sterilisation
     * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
     * Ovulation inhibitory progesterone-only pills (i.e., desogestrel)

   Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception

   Prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection
   * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days from the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
   * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence Male subjects must
   * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
   * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.

   All subjects must
   * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
   * Agree not to share study medication with another person and to return all unused study drug to the investigator.
9. Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
10. Able and willing to take heparin (usually low-molecular weight - LMWH) or low acetylsalicylic acid (100 mg) daily as prophylactic anticoagulation.
11. Life-expectancy > 3 months.

EXCLUSION CRITERIA

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Females, who are pregnant, calculate to get pregnant or are breast feeding (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Patient currently is enrolled in another clinical research study or has been enrolled in such a study within 4 weeks before randomization/registration and/or is receiving an investigational agent for any reason or has received such an agent within 4 weeks before randomization/registration.
5. Known hypersensitivity to thalidomide, dexamethasone, or cyclophosphamide or similar drugs.
6. Any prior use of lenalidomide.
7. Concurrent use of other anti-cancer agents or treatments.
8. Known positive for HIV or infectious hepatitis, type A, B or C.
9. Any other chemotherapy or high-dose dexamethasone within 4 weeks before randomization/registration.
10. Immunotherapy or antibody therapy within 8 weeks before randomization/registration.
11. Major surgery within 4 weeks before randomization/registration.
12. Myocardial infarction within 6 months before randomization/registration, New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
13. Cardiac amyloidosis.
14. Poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to the protocol.
15. Any systemic infection requiring treatment.
16. Cystitis.
17. Disturbance of urinary flow.
18. Unable or unwilling to take heparin (usually low-molecular weight - LMWH) or low acetylsalicylic acid (100 mg) daily as prophylactic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of CY (PO and IV) in combination with LEN/low-dose DEX | 3 years
To investigate the best objective response (EBMT criteria) to both treatment regimens | 3 years

SECONDARY OUTCOMES:
To investigate safety and tolerability of both treatment regimens | 3 years
To investigate other efficacy parameters of both treatment regimens | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kropff, MD, Study Chair — University of Münster, Department of Hematology/Oncology
Locations (4):
- Germany (4):
  - University Clinic München-Großhadern, München
  - University of Münster, Department of Hematology/Oncology, Münster
  - Tübingen University, Department of Hematology/Oncology/Immunology, Tübingen
  - University Clinic Ulm, Department Internal Medicine, Ulm